CLINICAL TRIAL: NCT05943457
Title: Efficacy of Vitamin K2 Supplementation in Adult Episodic Migraine
Brief Title: Vitamin K2 Supplementation in Adult Episodic Migraine
Acronym: ViKEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sola Aoun Bahous, M.D. Ph.D. (Other)
Collaborators: Lesaffre International (Industry); Omicron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Sola Aoun Bahous, M.D. Ph.D., Professor of Medicine, Lebanese American University
Organization: Lebanese American University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MK7-003
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Migraine Headache; Arterial Stiffness; Vitamin K Deficiency
Keywords: Migraine; Arterial stiffness; Vitamin K deficiency; Migraine attack
MeSH Terms: conditions — Migraine Disorders; Vitamin K Deficiency | interventions — Vitamin K 2; menaquinone 7

STUDY DESIGN:
Intervention Model Description: Migraine subjects will be randomized to receive either the supplement of vitamin K2 or a placebo for the duration of 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, investigators, and analysts will remain blind to the identity of the treatment from the time of randomization until the time of unblinding. The identity of the treatment will be concealed by using placebo pills that are identical in appearance, color, odor and packaging. Unblinding will only occur in the case of a medical emergency and at the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (MK7) Arm (Experimental): This corresponds to the sub-group of subjects who will receive the supplement (vitamin K2 or Menaquinone-7).
  Interventions: Dietary Supplement: Vitamin K2 or menaquinone-7
- Control Arm (Placebo Comparator): This corresponds to the sub-group of subjects who will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K2 or menaquinone-7 — Vitamin K2 (MK7) 360 mcg/day orally once daily for 6 months
  Other Names: MenaQ7
  Arms: Intervention (MK7) Arm
Other: Placebo — Placebo pills will be administered orally once daily for 6 months
  Arms: Control Arm

SUMMARY:
Migraine is a debilitating illness and a major cause of disability in the world. It is highly prevalent, especially among women. Vitamin supplementation is a potential therapeutic option for migraines that remains largely under-explored. Several studies have shown that people with migraine tend to have higher arterial stiffness than people without migraine. Vitamin K2 deficiency is an important mediator of arterial stiffness and calcification due to decreased carboxylation of matrix Gla protein (MGP). Supplementation reverses these changes and improves vascular health in patients with end stage renal disease according to previous studies. Therefore, vitamin K2 supplementation could serve a potential role in migraine patients. The purpose of the study is to test the effect of vitamin K2 on decreasing the frequency of migraine attacks and decreasing arterial stiffness. The population will be recruited from the neurology clinic at LAU Medical Center-Rizk Hospital and will constitute of adult patients. They will be randomized to receive either the supplement of vitamin K2 or a placebo for the duration of 6 months. Laboratory tests and arterial stiffness measurements will be done at the beginning, middle, and at the end of the study for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above
* History of episodic migraine with or without aura since > 12 months according to the ICHD-3 criteria.
* Migraine frequency from 4-14 days per month over the 3 months prior to screening.
* Migraine frequency from 4-14 days per month during the baseline period of assessment.
* Successful completion of the migraine diary during the baseline evaluation period.

Exclusion Criteria:

* Migraine patients with superimposed tension type or other forms of primary headaches
* Patients who are currently on any of the migraine prophylactic treatments (Sodium valproate, Topiramate, Beta-blockers, Tricyclic antidepressants, SRNI, Flunarizine, Verapamil, Lisinopril, Candesartan)
* Patients who have been on any of the previously listed medications within 3 months of screening
* Patient who takes the following medications:

  * Ergotamine or Triptans > 10 days per month
  * NSAIDs or paracetamol > 15 days per month
  * Opioids more than 4 days per month
  * Patients on anticoagulants
* Other active chronic pain syndromes (i.e. fibromyalgia, painful peripheral neuropathy, post-herpetic neuralgia…)
* History of hypersensitivity to the vitamin K2
* History of soy protein, cheese, eggs and meat allergy
* History of thrombotic events
* Diagnosed coagulopathy or any condition related to coagulation
* Cardiovascular event in the past month
* Current or planned pregnancy
* Lactation
* Inability to tolerate oral medications
* Known intestinal malabsorption or hypomotility syndromes
* Atrial fibrillation
* Active malignancy
* Any acute illness in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes of monthly migraine days | 6 months
  Effect of Vitamin K2 supplementation on the changes from baseline in monthly migraine days as compared to placebo. This will be assessed clinically using a questionnaire to be administered at the start, monthly, and at the end of the study (6 months) about frequency and number of migraine days per month.

SECONDARY OUTCOMES:
Changes from baseline in the headache impact score (HIT-6) as compared to placebo. | 6 months
Changes from baseline in monthly severe migraine days. | 6 months
  Changes from baseline in monthly severe migraine days as defined by a visual analogue scale rating above 7, as compared to placebo.
Changes from baseline on the modified migraine disability assessment (MIDAS) score as compared to placebo. | 6 months
Changes from baseline on the modified migraine physical function impact diary (MPFID) as compared to placebo. | 6 months
Changes from baseline on the quality of life as measure by the EuroQoL compared to placebo. | 6 months
Changes from baseline of arterial stiffness level. | 6 months
  Changes of arterial stiffness level assessed by measuring the cfPWV using Complior Analyze.

CONTACTS AND LOCATIONS:
Overall Officials: Sola Aoun Bahous, MD, PhD, Principal Investigator — Lebanese American University School of Medicine
Locations (1):
- Lebanese American University Medical Center - Rizk Hospital, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: We have a plan to publish the study protocol as soon as possible.

REFERENCES:
- [Background] Stovner Lj, Hagen K, Jensen R, Katsarava Z, Lipton R, Scher A, Steiner T, Zwart JA. The global burden of headache: a documentation of headache prevalence and disability worldwide. Cephalalgia. 2007 Mar;27(3):193-210. doi: 10.1111/j.1468-2982.2007.01288.x. PMID 17381554
- [Background] Kurth T, Winter AC, Eliassen AH, Dushkes R, Mukamal KJ, Rimm EB, Willett WC, Manson JE, Rexrode KM. Migraine and risk of cardiovascular disease in women: prospective cohort study. BMJ. 2016 May 31;353:i2610. doi: 10.1136/bmj.i2610. PMID 27247281
- [Background] Mozos I, Stoian D, Luca CT. Crosstalk between Vitamins A, B12, D, K, C, and E Status and Arterial Stiffness. Dis Markers. 2017;2017:8784971. doi: 10.1155/2017/8784971. Epub 2017 Jan 12. PMID 28167849
- [Background] Westenfeld R, Krueger T, Schlieper G, Cranenburg EC, Magdeleyns EJ, Heidenreich S, Holzmann S, Vermeer C, Jahnen-Dechent W, Ketteler M, Floege J, Schurgers LJ. Effect of vitamin K2 supplementation on functional vitamin K deficiency in hemodialysis patients: a randomized trial. Am J Kidney Dis. 2012 Feb;59(2):186-95. doi: 10.1053/j.ajkd.2011.10.041. Epub 2011 Dec 9. PMID 22169620
- [Background] Mansour AG, Hariri E, Daaboul Y, Korjian S, El Alam A, Protogerou AD, Kilany H, Karam A, Stephan A, Bahous SA. Vitamin K2 supplementation and arterial stiffness among renal transplant recipients-a single-arm, single-center clinical trial. J Am Soc Hypertens. 2017 Sep;11(9):589-597. doi: 10.1016/j.jash.2017.07.001. Epub 2017 Jul 13. PMID 28756183
- [Background] Mansour AG, Ahdab R, Daaboul Y, Korjian S, Morrison DA, Hariri E, Salem M, El Khoury C, Riachi N, Aoun Bahous S. Vitamin K2 Status and Arterial Stiffness Among Untreated Migraine Patients: A Case-Control Study. Headache. 2020 Mar;60(3):589-599. doi: 10.1111/head.13715. Epub 2019 Nov 25. PMID 31769041